CLINICAL TRIAL: NCT05835310
Title: A Phase III, Randomized, Double-blind, Parallel-group, Placebo Controlled Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy, and Safety of IV Anifrolumab in Pediatric Participants 5 to < 18 Years of Age With Moderate to Severe Active Systemic Lupus Erythematosus While on Background Standard of Care Therapy
Brief Title: An Efficacy and Safety Study of Intravenous Anifrolumab to Treat Systemic Lupus Erythematosus in Pediatric Participants
Acronym: BLOSSOM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3461C00030
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; Monoclonal Antibody; Anifrolumab; Parallel-group treatment; Pediatric participants; Standard of care therapy; Intravenous
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anifrolumab (Experimental): Randomized participants will receive anifrolumab via intravenous (IV) infusion every 4 weeks
  Interventions: Biological: Anifrolumab
- Placebo (Placebo Comparator): Randomized participants will receive matching placebo via IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Anifrolumab — Participants will receive anifrolumab via IV infusion.
  Other Names: (MEDI-546)
  Arms: Anifrolumab
Drug: Placebo — Participants will receive matching placebo via IV infusion
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Pharmacokinetics (PK), Pharmacodynamics (PD), Efficacy, and Safety of Anifrolumab in Children with Moderate to Severe Active Systemic Lupus Erythematosus (SLE)

DETAILED DESCRIPTION:
This study aims to characterize the pharmacokinetics, pharmacodynamics, efficacy, and safety of Anifrolumab solution for infusion compared with placebo solution for infusion in pediatric participants with severe active systemic lupus erythematosus who are on background standard of care therapy.

The study duration for a participant will be approximately 116 weeks, which includes:

* Screening period of up to 30 days.
* Part A consists of a four-week, double-blind, placebo-controlled, randomised, pharmacokinetic period.
* Part B is a double-blind, placebo-controlled, randomised, safety/efficacy period lasting 48 weeks (for rollover participants from Part A) or 52 weeks (for de novo participants).
* Part C is a 52-week open-label extension period.
* Part D is a safety follow-up period. One safety visit at 12 weeks post last dose.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent/caregiver/legally authorized representative and participant (if required per local country regulation) capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol. Informed assent is to be provided by the participant per local country regulation.
* Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) criteria for at least 3 months prior to signing the ICF.
* Participant should meet all of following tuberculosis (TB) criteria:

A. No signs or symptoms of active TB B. No medical history or past physical examinations suggestive of active TB C. No recent contact with a person with active TB or if there has been such contact, referral to a TB specialist for evaluation and initiation of treatment for latent TB, if warranted, prior to the first administration of study intervention in accordance with local SoC D. No history of latent TB without documented completion of treatment prior to initial screening visit

* Female participants of childbearing potential must have a negative serum pregnancy test at screening and negative urine pregnancy test at randomization.
* Female participants of childbearing and male participants must adhere to the contraception methods.
* At screening, negative SARS-CoV-2 RT-PCR or rapid antigen test result and no known or suspected COVID-19 infection or exposure between screening and randomization visits.

Exclusion Criteria:

* Known diagnosis of an IFN-mediated autoinflammatory interferonopathy.
* History of, or current diagnosis of, clinically significant non-SLE-related vasculitides.
* In participants aged 11 years and above: history or evidence of suicidal ideation.
* History of any non-SLE disease that has required treatment with oral or parenteral corticosteroids for more than a total of 2 weeks within the last 24 weeks prior to signing the ICF.
* Any positive result on screening for human immunodeficiency virus.
* Active hepatitis B surface antigen OR hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody and detectable HCV ribonucleic acid (RNA) or any active or recent case of Herpes Zoster infection.
* Any clinical cytomegalovirus or Epstein-Barr virus infection that has not completely resolved within 12 weeks prior to signing the ICF.
* History of severe COVID-19 infection requiring hospitalization, intensive care unit care, or assisted ventilation or any prior COVID-19 infection with unresolved sequelae. Any mild/asymptomatic COVID-19 infection (laboratory confirmed or suspected based on clinical symptoms).
* Prior use of anifrolumab.
* Prior treatment with directly acting cytotoxic B-cell depleting therapeutics (eg, rituximab) < 26 weeks prior to ICF signature.
* Blood transfusion or receipt of blood products except albumin within 4 weeks prior to signing the ICF.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2028-10-05 (Estimated); Study Completion 2030-01-09 (Estimated)

PRIMARY OUTCOMES:
Part A- Anifrolumab serum concentration | Up to Day 29
  The serum concentration will be characterised and the dose of anifrolumab will be defined in pediatric participants with moderate to severely active SLE.
Part A - Maximum observed serum (peak) drug concentration (Cmax) | Up to Day 29
  The serum PK will be characterised and the dose of anifrolumab will be defined in pediatric participants with moderate to severely active SLE.
Part A - Area under the serum concentration curve (AUC) | Up to Day 29
  The serum PK will be characterised and the dose of anifrolumab will be defined in pediatric participants with moderate to severe active SLE.
Part A - Minimum observed serum concentration (Cmin) | Up to Day 29
  The serum PK will be characterised and the dose of anifrolumab will be defined in pediatric participants with moderate to severe active SLE.
Part B - Number of participants who are British Isles Lupus Assessment Group-based Composite Lupus Assessment (BICLA) responders (yes/no) | At Week 52
  BICLA response is defined as:
  * Reduction of all baseline British Isles Lupus Assessment Group BILAG-2004 A to B/C/D and B to C/D, and no BILAG-2004 worsening in other organ systems, as defined by ≥ 1 new BILAG-2004 A or ≥ 2 new BILAG- 2004 B.
  * No worsening from baseline in SLEDAI-2K, defined as an increase from baseline of > 0 points.
  * No worsening from baseline in participant's lupus disease activity, defined by an increase ≥ 0.30 points on a PGA 3-point visual analogue scale (VAS).

SECONDARY OUTCOMES:
Part B - Number of participants who are Systemic Lupus Erythematosus Responder Index of ≥ 4 SRI(4) responders (yes/no) | At Week 52
  SRI-4 response is defined as:
  * ≥ 4-point reduction from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score.
  * No new organ systems affected as defined by ≥ 1 new BILAG-2004 A or ≥ 2 new BILAG-2004 B items compared to baseline.
  * No worsening from baseline in participant's lupus disease activity, defined by an increase ≥ 0.30 points on a PGA 3-point VAS.
Part B - Time to first flare | Through Week 52
  Time to first flare, where flare is defined as either ≥ 1 new BILAG-2004 A, or ≥ 2 new BILAG-2004 B items compared with the previous visit.
Part - B Change from baseline through Week 52 in anifrolumab serum concentration | Baseline, Week 52
  The PK of anifrolumab in pediatric participants with moderate to severe active SLE will be characterized.
Part - B Change from baseline through Week 52 in antidrug antibody (ADA) | Baseline, Week 52
  The immunogenicity of anifrolumab in pediatric participants with moderate to severe active SLE will be characterized.
Part - B Change from baseline in anti-double stranded deoxyribonucleic acid antibodies | Baseline, Week 52
  The PD of anifrolumab in pediatric participants with moderate to severe active SLE will be characterized.
Part - B Change from baseline through Week 52 in complement components and CH50 | Baseline, Week 52
  The PD of anifrolumab in pediatric participants with moderate to severe active SLE will be characterized.
Number of participants who are Pediatric Rheumatology International Trials Organization/American College of Rheumatology (PRINTO/ACR) childhood-onset systemic lupus erythematosus (cSLE) responders (yes/no) | At Week 52
  PRINTO/ACR cSLE responders are defined as participants with at least 50% improvement from baseline in any 2 of 5 core set outcome measures and no more than one of the remaining worsening more than 30%, where the core set measures are:
  * ParentGA 21-circle VAS
  * PGA 3-point VAS
  * SLEDAI-2K
  * PedsQL Generic Core (Physical Functioning Domain)
  * Proteinuria
Part B - The mean percentage reduction from Baseline through Week 52 in oral corticosteroid(s) (OCS) background dose | Baseline, Week 52
  The efficacy of anifrolumab vs placebo on OCS background dose in pediatric participants with moderate to severe active SLE will be characterized.
Part B - Change from baseline through Week 52 in type I interferon (IFN) 21-gene signature | Baseline, Week 52
  Type 1 IFN 21 gene signatures in pediatric patients with moderate to active SLE will be characterized.

OTHER OUTCOMES:
All parts - Number of participants reporting suicidal ideation and/or suicidal behavior as per Columbia Suicide Severity Rating Scale (C-SSRS) | From Week 0 until the follow-up visit (12 weeks post-last dose)
  The safety and tolerability of anifrolumab in pediatric participants with moderate to severe active SLE will be assessed.
All parts - Number of participants with adverse events | From Week 0 until the follow-up visit (12 weeks post-last dose)
  The safety and tolerability of anifrolumab in pediatric participants with moderate to severe active SLE will be assessed.

CONTACTS AND LOCATIONS:
Locations (86):
- United States (21):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Saint Paul, Minnesota
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
- Argentina (3):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Rosario
- Brazil (5):
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, São Paulo
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- China (7):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Wenzhou
  - Research Site, Zhengzhou
- Colombia (2):
  - Research Site, Barranquilla
  - Research Site, Medellín
- France (5):
  - Research Site, Bordeaux
  - Research Site, Bron
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Lille
  - Research Site, Toulouse
- Germany (3):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Sankt Augustin
- Italy (4):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Japan (8):
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fuchu-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Obu-shi
  - Research Site, Shinjuku-ku
  - Research Site, Yokohama
- Mexico (5):
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Toluca
- Poland (3):
  - Research Site, Lodź
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Research Site, Cape Town, South Africa
- Spain (4):
  - Research Site, Esplugues de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Kayseri
  - Research Site, Umraniye
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patientlevel data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home